CLINICAL TRIAL: NCT01718756
Title: Efficacy of Continuous Intravenous Infusion vs. Scheduled Dosing of Lornoxicam on Patient Controlled Morphine Consumption After Orthopaedic Surgery: A Comparative Placebo Study
Brief Title: Continuous Lornoxicam Infusion for Orthopaedic Surgery
Status: Suspended | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: No enough fund or cases
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Mohamed R El Tahan, Associate Professor of Anesthesiology & SICU, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R/55
Record Dates: First submitted 2012-10-28; First posted 2012-10-31 (Estimated); Last update posted 2020-09-04 (Actual); Status verified 2020-09

CONDITIONS: Closed Non Comminuted Long Bone Fractures
Keywords: Orthopaedic; General anaesthesia; lornoxicam; patient controlled analgesia; morphine consumption
MeSH Terms: interventions — Appointments and Schedules

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator): The placebo group received 12 hourly boluses of 0.9% saline, followed by a constant infusion for 48 hrs after surgery.
  Interventions: Drug: Placebo
- Scheduled (Active Comparator): They received a 12 hourly boluses of lornoxicam followed by a constant infusion of 0.9% saline, for 48 hrs after surgery
  Interventions: Drug: Scheduled
- Continuous infusion (Active Comparator): They received boluses of lornoxicam 0.8 mg/mL before induction of anaesthesia followed by a 12 hourly boluses of 0.9% saline and a constant infusion at 10 mL/h of lornoxicam 0.13 mg/mL, for 48 hrs. after surgery.
  Interventions: Drug: Continuous infusion

INTERVENTIONS:
Drug: Placebo — The placebo group received 12 hourly 20-mL i.v. boluses of 0.9% saline starting 20 min before induction of anaesthesia, followed by a constant infusion at 10 mL/h, for 48 hrs after surgery.
  Arms: Placebo
Drug: Continuous infusion — The "continuous infusion" group received 20-mL i.v. boluses of lornoxicam 0.8 mg/mL starting 20 min before induction of anaesthesia followed by a 12 hourly 20-mL i.v. boluses of 0.9% saline and a constant infusion at 10 mL/h of lornoxicam 0.13 mg/mL, for 48 hrs. after surgery
  Arms: Continuous infusion
Drug: Scheduled — The "scheduled" group received an 12 hourly 20-mL i.v. boluses of lornoxicam 0.8 mg/mL starting 20 min before induction of anaesthesia followed by a constant infusion at 10 mL/h of 0.9% saline, for 48 hrs after surgery (supplied by Xefo, JPI, Saudi Arabia), starting 20 min before induction of anaesthesia.
  Arms: Scheduled

SUMMARY:
Perioperative continuous infusion of lornoxicam would be an effective and safe regimen to reduce the patient controlled morphine consumption after orthopaedic surgery.

After ethical approval, 96 patients scheduled for elective orthopaedic fracture surgery under general anaesthesia were randomly allocated to receive placebo, 12-hourly iv lornoxicam 16 mg or lornoxicam 16 mg followed with continuous infusion of 1.3 mg/hr., for 48 hours after surgery (n=32 per group). Anaesthesia was induced with propofol, sufentanil and rocuronium, and was maintained with 0.5-1 minimum alveolar concentration sevoflurane, sufentanil and rocuronium. Postoperative patient controlled morphine analgesia was used. Changes in heart rate, mean blood pressure and sevoflurane minimum alveolar concentration, visual analogue pain scores, and cumulative patient controlled morphine consumptions and blood loss for 48 hours, platelet functions, bone non-union and the presence of adverse effects were recorded.

DETAILED DESCRIPTION:
An independent investigator who was not involved in the study instructed the patients preoperatively about the use of visual analogue scale to assess the severity of postoperative pain (0 mm for no pain and100 mm for worst imaginable pain) and about the use of PCA for their postoperative pain management.

Anaesthetic management was standardized. Oral lorazepam 2 mg was given the night before surgery. Subjects were allocated randomly into three groups (n = 32 for each) by drawing sequentially numbered sealed opaque envelopes containing a software-generated randomization code (Random Allocation Software, version 1.0.0, Isfahan University of Medical Sciences, Isfahan, Iran)into the placebo, scheduled, and continuous infusion groups. The syringes containing placebo and lornoxicam solutions were masked by identical opaque identical cover sheets. The test solution was prepared by one anaesthesiologist before induction of anaesthesia. Another anaesthesiologist, who was blinded to the study solution, gave the anaesthetic and was instructed to avoid using local anaesthetics, and a third anaesthesiologist collected perioperative data. All staff in the operating room were unaware of patient allocation group.

Patient monitoring included electrocardiography, non-invasive blood pressure, pulse oximetry, end-tidal sevoflurane and carbon dioxide (ETCO2) concentrations, response entropy (RE) and state entropy (SE.

After preoxygenation for 3 min, anesthesia was induced with fentanyl 1 - 3 µg/kg, propofol 1.5-2.5 mg/kg (to achieve an SE <50 and a difference<10 between RE and SE; RE-SE) and rocuronium 0.6 mg/kg. Tracheal intubation or slipping of laryngeal mask appropriate for body weight were used according to the discretion of the attending anaesthetist. Anaesthesia was maintained with a 0.6-1 minimum alveolar concentration of sevoflurane (MAC-Sevo) with air in 40% oxygen and fentanyl 1 µg/kg boluses to maintain SE <50 and RE-SE <10 and heart rate and mean arterial blood pressure within 20% of their baseline values. Rocuronium 0.1 mg/kg was given to maintain suppression of the second twitch using a train-of-four stimulation. The patients' lungs were ventilated to maintain an ETCO2 of 30-35 mmHg. Sevoflurane were discontinued at the start of skin closure, residual neuromuscular block was antagonized and the trachea extubated.

Postoperative analgesia was achieved according to the hospital protocol with patient controlled morphine analgesia (1 mg/ml), 1 mg, with a lockout interval of 8 minutes and a maximum 24-hourly limit of 180 mg. respiratory depression defined as the decrease in respiratory rate below 8/min was treated with i.v naloxone 0.2 mg. Nausea and vomiting were treated with i.v granisetron 1 mg and pruritus was treated with i.m promethazine 25 mg.

Heart rate and mean arterial blood pressure were recorded before (baseline) and 10 min after the start of infusion; every 30 min during surgery; every 15 min during the stay in post anaesthesia care unit (PACU), and 8 hourly for the following 48 hours. MAC-Sevo was recorded every 15 min after intubation until the end of surgery. Intraoperative fentanyl consumption was recorded.

The VAS pain scores, the presence and intensity of postoperative sedation (four-point verbal rating scores (VRS): awake, drowsy, rousable or deep sleep), nausea and vomiting (0: no nausea; 1: nausea no vomiting; 2: nausea and vomiting), were reported every 15 min for the first postoperative hour and two-hourly thereafter for the first 48 postoperative hours. The cumulative morphine consumption during the first 24 and 48 postoperative hours were recorded.

Platelet function assay was performed before and every 24 hrs. for the first three days after surgery. Cumulative intraoperative and postoperative blood loss and the number of transfused blood units were recorded. The presence of fracture non-union was reported.

All patients were observed by an independent investigator during the study period for the presence of nausea, vomiting, gastritis, reflux esophagitis, headache, bleeding, bronchospasm, sweating, allergy, thrombocytopenia, bleeding, ecchymosis, or increases in liver transaminases.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists physical class I to III
* Age from 18 to 55 years
* Closed non comminuted long bone fractures
* Elective orthopaedic fracture surgery
* General anaesthesia

Exclusion Criteria:

* Hypersensitivity to lornoxicam
* Gastrointestinal ulceration or bleeding
* Cardiac diseases
* Pulmonary diseases
* Hepatic diseases
* Renal diseases
* Clotting diseases
* Bleeding diseases
* Bronchial asthma
* Diabetes mellitus
* Peripheral arterial occlusive disease
* Morbid obesity
* Pregnancy
* Alcohol or drug abuse
* Receiving other NSAIDs a day before surgery

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 96 (Estimated)
Dates: Start 2013-06 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
postoperative patient controlled morphine consumption | 24 hours and 48 hours after surgery
  The cumulative morphine consumption during the first 24 and 48 postoperative hours were recorded.

SECONDARY OUTCOMES:
Quality of analgesia | every two hours for 24 hours after surgery
  the use of visual analogue scale to assess the severity of postoperative pain (0 mm for no pain and100 mm for worst imaginable pain)
platelet functions | daily after surgery for three days
Bone non-union | for 3 months after surgery
postoperative sedation | every two hours for 24 hours after surgery
  four-point verbal rating scores (VRS): awake, drowsy, rousable or deep sleep),
Nausea and vomiting | every two hours for 24 hours after surgery
  nausea and vomiting (0: no nausea; 1: nausea no vomiting; 2: nausea and vomiting),
Perioperative blood loss | Cumulative intraoperative and 24 hours after surgery

OTHER OUTCOMES:
Lornoxicam adverse effects | 48 hours after surgery
  the presence of nausea, vomiting, gastritis, reflux esophagitis, headache, bleeding, bronchospasm, sweating, allergy, thrombocytopenia, bleeding, ecchymosis, or increases in liver transaminases.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed R El Tahan, MD, Principal Investigator — College of Medicine, Mansoura University
Locations (1):
- Anesthesiology Dept., College of Medicine, Mansoura University, Al Mansurah, DK, Egypt